CLINICAL TRIAL: NCT04126616
Title: Pulmonary Vascular Impairment in Chronic Obstructive Pulmonary Disease (COPD) Assessed by MRI
Acronym: PulmoVasc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-14
Record Dates: First submitted 2019-10-09; First posted 2019-10-15 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with COPD and PH (Experimental)
  Interventions: Diagnostic Test: chest Magnetic Resonance Imaging (MRI) using Gadolinium-based contrast agent
- patients with COPD without PH (Active Comparator)
  Interventions: Diagnostic Test: chest Magnetic Resonance Imaging (MRI) using Gadolinium-based contrast agent
- healthy subjects (Active Comparator)
  Interventions: Diagnostic Test: chest Magnetic Resonance Imaging (MRI) using Gadolinium-based contrast agent

INTERVENTIONS:
Diagnostic Test: chest Magnetic Resonance Imaging (MRI) using Gadolinium-based contrast agent — chest MRI will be performed at rest and after moderate exercise

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a highly prevalent pulmonary disease providing major morbidity and mortality. Bronchial obstruction is the cornerstone in assessment of the disease whereas associated pulmonary vascular disease remains poorly known.

Improving knowledge on pulmonary vascular adaptive skills in COPD patients could allow for better understanding disease exacerbations, evolution towards chronic pulmonary hypertension (PH) and therapeutics to be offered to the patients.

Magnetic resonance imaging (MRI) is an innovative and non-invasive tool capable of pulmonary vascular evaluation. This work aims at identifying pulmonary vascular impairment in COPD patients using functional MRI.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a highly prevalent pulmonary disease providing major morbidity and mortality. Bronchial obstruction is the cornerstone in assessment of the disease whereas associated pulmonary vascular disease remains poorly known.

However, it has been shown that emphysema, frequently observed in COPD, contains major vascular lesions. Alteration of pulmonary vascularisation have been found during exacerbation of the disease.

Moreover, it is well established that such vascular lesions form the substrate for endothelial dysfunction, expressed as an impairment of vascular adaptation during exercise, and evolving towards chronic pulmonary hypertension (PH). Owing to its severe effects on the right-sided heart, it signs a pejorative turn in patients' survival and quality of life.

Finally, COPD patients' phenotypes are very heterogeneous and the clinical response to PH treatments is variable; while some get a benefit, others are counter-indicated due to adverse effects.

Improving knowledge on pulmonary vascular adaptive skills in COPD patients could allow for better understanding disease exacerbations, evolution towards PH and therapeutics to be offered to the patients.

This area of research remains widely unknown because of the lack of simple tools to assess pulmonary vascularisation which could be used in clinical routine. Magnetic resonance imaging (MRI) is an innovative and non-invasive tool capable of pulmonary vascular evaluation. This work aims at identifying pulmonary vascular impairment in COPD patients using functional MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Diagnosed with COPD
* Emphysema on chest CT
* FEV1 between 35 and 80 %
* Screened for PH by echocardiography

Exclusion Criteria:

* side effect for exercise
* side effect for MRI and contrast agent injection
* Pregnancy or breastfeeding
* Refusing to be informed of the discovery of an anomaly on chest MRI

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Pulmonary blood flow variation from rest to exercise | 4 hours
  Pulmonary blood flow will be measured with dynamic contrast-enhancement MRI at rest and after moderate exercise. Relative variation is the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France